CLINICAL TRIAL: NCT04954521
Title: A Real World Study on the Effect of Single or Combined Treatment of Anlotinib on Survival and Prognosis of Advanced Hepatocellular Carcinoma
Brief Title: Anlotinib for Hepatocellular Carcinoma
Acronym: AFHC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: People's Hospital of Guangxi Zhuang Autonomous Region (Other)
Responsible Party: Principal Investigator, Kehe Chen, Chief physician, People's Hospital of Guangxi Zhuang Autonomous Region
Other Study IDs: KY-QT-201905
Record Dates: First submitted 2021-06-17; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Liver Neoplasms
MeSH Terms: conditions — Liver Neoplasms | interventions — anlotinib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Anlotinib — This is an observational study

SUMMARY:
The purpose of this study is to observe and explore the effect of single or combined treatment of arotinib on the survival and prognosis of patients with advanced liver cancer in the real world, and to summarize the treatment experience of a wide range of people.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 18 years old, male or female;
2. Patients with advanced liver cancer were diagnosed;
3. Patients assessed by doctors to benefit from single or combined treatment of arotinib;
4. Patients volunteered to join the project.

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with advanced liver cancer
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-06-30 (Estimated); Primary Completion 2023-07-05 (Estimated); Study Completion 2024-07-05 (Estimated)

PRIMARY OUTCOMES:
OS | From date of admission until the date of death from any cause, assessed up to 24 months
  Overall Survival

SECONDARY OUTCOMES:
PFS | From date of admission until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Progression Free Survival

CONTACTS AND LOCATIONS:
Locations (1):
- People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: No